CLINICAL TRIAL: NCT05581069
Title: Improving Outcomes in Autism: Community Implementation of Stepped Transition in Education Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alabama, Tuscaloosa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A22-0209
Record Dates: First submitted 2022-09-29; First posted 2022-10-14 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; adult; transition; employment
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: This is a single-arm (non-randomized) trial in which providers are community-based practitioners.
Masking Description: The assessment battery is multi-modal and includes evaluation by an independent evaluator (IE) who is uninvolved in STEPS delivery or training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STEPS (Experimental): All participants receive the STEPS intervention
  Interventions: Behavioral: STEPS

INTERVENTIONS:
Behavioral: STEPS — STEPS is a psychosocial intervention that targets self-determination, self-regulation, and self-knowledge to improve functional independence and quality of life in adults.

SUMMARY:
The goal of this study is to conduct the first community-based implementation of the STEPS program and test feasibility and preliminary impact. After first working with stakeholders to refine and optimize the program we will launch a Hybrid Type 1 open trial, targeting 25 transition-age youth (TAY) with ASD.

DETAILED DESCRIPTION:
This community-engaged, applied research study will test the effectiveness of STEPS (Stepped Transition in Education Program for Students with ASD), a program designed to help transition-age youth (TAY) with ASD prepare for independence. Adults with ASD have worse outcomes, with respect to employment, education, and quality of life, than neurotypical peers. Research-informed transition planning that addresses core impairments in skills needed for autonomous and independent living, including self-knowledge, self-determination, and self-regulation, may improve outcomes for this growing population. In a prior trial, the investigators found STEPS to be feasible, acceptable, and efficacious. The proposed study is the first test of STEPS as implemented by community-based providers. Through a series of implementation working group meetings with identified community partner agency and stakeholders (families, TAY with ASD) in the region, the study team will refine STEPS with the goal of optimizing program sustainability within community settings. Following this, a Hybrid Type 1 open trial will be launched, which focuses primarily on intervention effectiveness with a secondary focus on factors related to implementation. With a sample of TAY with ASD (n=25) immediate and longer-term clinical outcomes of adult functional outcomes and vocational engagement will be assessed. This research will produce findings with the potential to shift clinical practice related to transition to adulthood for people with ASD.

ELIGIBILITY:
Inclusion Criteria:

* ages 16-25 confirmed diagnosis of ASD caregiver willing to participate stable medication

Exclusion Criteria:

* evidence of intellectual disability evidence of suicidal intent

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Adult Functioning Scale | Week 14
  The Adult Functioning Scale measures autonomy, employment (including readiness), social functioning, and satisfaction via self- and informant-report questionnaires
Rehabilitation Success | Week 14
  This is completed via interview to assess 'real world' vocational engagement

CONTACTS AND LOCATIONS:
Overall Officials: Susan W White, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Center for Youth Development and Intervention, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
There is no pre-existing plan, but de-identified data will be shared after publication of main findings, upon request.

REFERENCES:
- [Background] White SW, Smith IC, Miyazaki Y, Conner CM, Elias R, Capriola-Hall NN. Improving Transition to Adulthood for Students with Autism: A Randomized Controlled Trial of STEPS. J Clin Child Adolesc Psychol. 2021 Mar-Apr;50(2):187-201. doi: 10.1080/15374416.2019.1669157. Epub 2019 Oct 14. PMID 31609666
- [Background] Elias R, White SW. Autism Goes to College: Understanding the Needs of a Student Population on the Rise. J Autism Dev Disord. 2018 Mar;48(3):732-746. doi: 10.1007/s10803-017-3075-7. PMID 28255760
- [Background] White SW, Elias R, Capriola-Hall NN, Smith IC, Conner CM, Asselin SB, Howlin P, Getzel EE, Mazefsky CA. Development of a College Transition and Support Program for Students with Autism Spectrum Disorder. J Autism Dev Disord. 2017 Oct;47(10):3072-3078. doi: 10.1007/s10803-017-3236-8. PMID 28685409